CLINICAL TRIAL: NCT07105930
Title: A Randomized Controlled Multicentric Trial to Assess Non-inferiority of an Orbital Atherectomy Only Versus a Calcium-tailored Debulking Approach
Brief Title: Trial to Assess Non-inferiority of an Orbital Atherectomy Only Versus a Calcium-tailored Debulking Approach
Acronym: OrFitA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDR-005
Record Dates: First submitted 2025-07-25; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Orbital Atherectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Debulging with the orbital atherectomy system (Diamondback 360®) (Experimental)
  Interventions: Device: Debulging approach using the orbital atherectomy system
- Debulging with various available methods (Active Comparator)
  Interventions: Procedure: Debulging using rotational atherectomy, scoring or cutting balloons, or shockwave therapy

INTERVENTIONS:
Device: Debulging approach using the orbital atherectomy system — A uniform approach using only the orbital atherectomy system (Diamondback 360®), which sands away the calcium with a rotating crown
  Arms: Debulging with the orbital atherectomy system (Diamondback 360®)
Procedure: Debulging using rotational atherectomy, scoring or cutting balloons, or shockwave therapy — A tailored approach, where the operator chooses from various available methods based on the patient's specific type of calcium
  Arms: Debulging with various available methods

SUMMARY:
Some patients with coronary artery disease have severely calcified vessels. In these cases, placing a stent - a small tube that helps keep the artery open - can be very difficult. Calcium build-up in the artery wall may prevent the stent from expanding properly, increasing the risk of complications or failure of the treatment.

To prepare these vessels before stenting, doctors use special techniques to modify or remove the calcium. These techniques are known as plaque modification strategies and can include devices such as atherectomy systems, scoring balloons, or intravascular lithotripsy. However, there is no clear standard as to which strategy is best.

Purpose of the Study:

This study compares two different approaches to treating calcified coronary arteries before stenting:

* A uniform approach using only the orbital atherectomy system (Diamondback 360®, Abbott), which sands away the calcium with a rotating crown
* A tailored approach, where the operator chooses from various available methods (e.g., rotational atherectomy, scoring or cutting balloons, or shockwave therapy) based on the patient's specific type of calcium The goal is to determine whether the uniform orbital atherectomy approach is not worse (non-inferior) than the individualized method when it comes to how well the stent expands inside the artery.

This is a randomized, controlled clinical trial. Patients will be randomly assigned to one of the two groups.

Randomization ensures fair comparison between both groups. The decision to implant a stent and to use additional techniques is at the discretion of the interventional cardiologist.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* Chronic coronary syndrome with a clinical indication for percutaneous coronary intervention of a severely calcified lesion as defined by coronary computer tomography (CT; Agatston Score of target lesion ≥453 OR Calcium Arc >270°). The determination of calcification in the target lesion is based on native and contrast enhanced CT scans that are conducted as per clinical guidelines. The CT images must not be older than 6 months at the time of patient enrollment.
* Signed informed consent
* The patient is an appropriate candidate for bypass surgery, angioplasty, or atherectomy therapy

Exclusion Criteria:

* Acute ST-Elevation Acute Coronary Syndrome (STE-ACS) within 48 hours
* Cardiogenic shock
* Chronic total occlusion of the target lesion
* Glomerular filtration rate < 30 ml/min/1.73 m2
* Known presence, at the time of enrollment, of any contraindications listed in the Instructions for Use (IFU) of the investigational device:

  * The OCT (optical coherence tomography) imaging catheter cannot cross
  * The wire or imaging catheter cannot cross
  * The target lesion is within a bypass graft or stent
  * The patient is not an appropriate candidate for bypass surgery, angioplasty, or atherectomy therapy.
  * The patient has angiographic evidence of thrombus
  * The patient has only one open coronary vessel
  * The patient has angiographic evidence of flow reducing dissection at the treatment site
  * The patient has a known hypersensitivity to egg-, soy-, or peanut protein or to any of the active substances or excipients of the ViperSlide™ lubricant
  * Pregnancy (assessed by clinical routine testing)
* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Post-procedural Minimal Stent Area (MSA %) as assessed by optical coherence to-mography (OCT) imaging | MSA will be assessed in the final OCT run performed after stent implantation withine baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ochs, PD Dr., Principal Investigator — Universitäres Herz- und Gefäßzentrum Frankfurt ZIM - Med. Clinic 3 - Cardiology and Angiology